CLINICAL TRIAL: NCT01342718
Title: Effect of Herbal Extract Granules Combined With Probiotics on Irritable Bowel Syndrome With Diarrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Seok-Jae Ko, Resident, Department of Internal Medicine, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2010-011
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Herbal medicine; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GJS/Duolac7S (Experimental): GJS: Real herbal extract granule/Duolac7S: Real probiotics
  Interventions: Dietary Supplement: Herbal extract granule and probiotics
- GJS-P/Duolac7S (Placebo Comparator): GJS-P: Placebo herbal extract granule/Duolac7S: Real probiotics
  Interventions: Dietary Supplement: Placebo herbal extract granule and probiotics
- GJS/Duolac7S-P (Placebo Comparator): GJS: Real herbal extract granule/Duolac7S-P: Placebo probiotics
  Interventions: Dietary Supplement: Herbal extract granule and placebo probiotics
- GJS-P/Duolac7S-P (Placebo Comparator): GJS-P: Placebo herbal extract granule/Duolac7S-P: Placebo probiotics
  Interventions: Dietary Supplement: Placebo herbal extract granule and placebo probiotics

INTERVENTIONS:
Dietary Supplement: Herbal extract granule and probiotics — The herbal extract granule, Gwakhyangjeonggisan granule, consists of 11 herbs. Ingredients: Agastachis, Perillae Folium, Angelicae Radix, Arecae Pericarpium, Hoelen, Magnoliae officinalis Cortex, Atractylis Rhizoma, Aurantii nobilis Percarpium, Pinelliae Rhizoma, Platycodi Radix, Glychrrhizae Radix. Dosage and frequency: 1 pack (3g), 3 packs per day (2 hours after morning, afternoon and evening meal)
  The probiotics, Duolac7S, consist of 7 bacteria. Ingredients: Lactobacillus acidophilus, L. plantarum, L. rhamnosus, Bifidobacterium breve, B. lactis, B. longum, Streptococcus thermophilus. Dosage and frequency: 1 capsule (5✕1,000,000,000 bacteria/capsule [7✕100,000,000 viable cells/strain]), 2 capsules per day (2 hours after morning and evening meal)
  Other Names: Gwakhyangjeonggisan granule and Duolac7S
  Arms: GJS/Duolac7S
Dietary Supplement: Herbal extract granule and placebo probiotics — The herbal extract granule, Gwakhyangjeonggisan granule, consists of 11 herbs. Ingredients: Agastachis, Perillae Folium, Angelicae Radix, Arecae Pericarpium, Hoelen, Magnoliae officinalis Cortex, Atractylis Rhizoma, Aurantii nobilis Percarpium, Pinelliae Rhizoma, Platycodi Radix, Glychrrhizae Radix. Dosage and frequency: 1 pack (3g), 3 packs per day (2 hours after morning, afternoon and evening meal).
  Duolac7S placebo has the same form, color and flavor as experimental intervention (Duolac7S). The dosage, frequency and duration is also the same as experimental intervention (Duolac7S).
  Other Names: Gwakhyangjeonggisan granule and placebo Duolac7S
  Arms: GJS/Duolac7S-P
Dietary Supplement: Placebo herbal extract granule and probiotics — The Gwakhyangjeonggisan placebo has the same form, color and flavor as experimental intervention (Gwakhyangjeonggisan). The dosage, frequency and duration is also the same as experimental intervention (Gwakhyangjeonggisan).
  The probiotics, Duolac7S, consist of 7 bacteria. Ingredients: Lactobacillus acidophilus, L. plantarum, L. rhamnosus, Bifidobacterium breve, B. lactis, B. longum, Streptococcus thermophilus. Dosage and frequency: 1 capsule (5✕1,000,000,000 bacteria/capsule [7✕100,000,000 viable cells/strain]), 2 capsules per day (2 hours after morning and evening meal)
  Other Names: Placebo Gwakhyangjeonggisan granule and Duolac7S
  Arms: GJS-P/Duolac7S
Dietary Supplement: Placebo herbal extract granule and placebo probiotics — The Gwakhyangjeonggisan placebo has the same form, color and flavor as experimental intervention (Gwakhyangjeonggisan). The dosage, frequency and duration is also the same as experimental intervention (Gwakhyangjeonggisan).
  Duolac7S placebo has the same form, color and flavor as experimental intervention (Duolac7S). The dosage, frequency and duration is also the same as experimental intervention (Duolac7S).
  Other Names: Placebo Gwakhyangjeonggisan granule and placebo Duolac7S
  Arms: GJS-P/Duolac7S-P

SUMMARY:
The aims of this study are to investigate the effect of famous herbal formula extract and probiotics on irritable bowel syndrome with diarrhea, and to determine whether these two experimental items affect intestinal permeability and the composition of intestinal microbiota.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS), a common chronic gastrointestinal disorder characterized by abdominal pain and alteration of bowel habits in the absence of structural abnormality, has a prevalence of approximately 15% in western populations1,2. Patients with IBS can be classified by their predominant bowel habits: diarrhea-predominant IBS (D-IBS), constipation-predominant IBS, or IBS with alternating bowel movements3. Although smooth-muscle relaxants, bulking agents, and anti-diarrheal agents are commonly used as conventional IBS treatments, many IBS patients turn to alternative treatments because of the lack of therapeutic advantages of these treatments4. Therefore, the development of a new therapy is necessary for IBS patients.

Gwakhyangjeonggisan (GJS; Kkako-shoki-san in Kampo Medicine; Huoxiang-zhengqi-san in Traditional Chinese Medicine), which was recorded originally in the famous ancient herbal formula literature "Formularies of the Bureau of people's Welfare Pharmacies", consists of 13 common crude herbs. GJS contains the chemical ingredients naringin, hesperidin, thymol, honokiol and magnolol5. GJS has been shown to protect intestinal barrier function6, contract the colonic muscle7, and regulate infectious diarrhea8 in vivo. In traditional Korean medicine, this herbal formula has long been used for relieving abdominal pain, diarrhea, and vomiting as an over-the-counter or prescribed medicine9-11. However, there have been no clinical trials to investigate the efficacy of GJS in IBS.

Probiotics are defined as viable microorganisms, which confer potential health benefits on the host when taken in proper amounts12. They are easily available, do not require a prescription, and are administered extensively for the relief of abdominal symptoms13. According to a recent systematic review and meta-analysis study, probiotics caused a modest improvement in the overall IBS symptoms14. The rationale for using probiotics for IBS is based on the assumption that they modify the composition of the intestinal microflora15 and regulate intestinal permeability by modulating the epithelial tight junctions16. Duolac7S (DUO), a probiotic mixture, contains 7 bacterial species including Bifidobacterium, Lactobacillus, and Streptococcus. Each of these bacterial species is reportedly beneficial for IBS17. DUO has been approved by the Korean Food and Drug Administration for restoring the ecological balance of intestinal microflora and improving intestinal symptoms18. Although DUO has been widely used as an over-the-counter product for IBS-related symptoms, no clinical trials have investigated the efficacy of DUO on IBS.

Recently, several herbal formulas and probiotics have been simultaneously administered to IBS patients for relieving abdominal symptoms19. In addition to lack of clinical evidence for the use of GJS or DUO, the efficacy of their combined treatment for IBS has not been elucidated. Thus, there is a need to evaluate the safety and efficacy of administration of GJS, DUO, or a combination therapy as a frequently used treatment for IBS. In the current trial, we identified the safety and efficacy of GJS, DUO, or a combination therapy on D-IBS by evaluating IBS symptoms and quality of life. To investigate their mechanisms in humans, intestinal permeability and composition of intestinal microbiota were assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 75, with a elementary-school diploma or higher, must be literate
2. One who meet Rome Ⅲ IBS-D criteria
3. One who agree on not taking other therapies during experimental period
4. During the past 5 yrs, no history of organic lesion proven by colonoscopy
5. One who agree on consent form

Exclusion Criteria:

1. Patients who have abdominal operation in the past(exception: appendectomy, caesarean section, tubal ligation, laparoscopic cholecystectomy, hysterectomy and abdominal wall hernia repair)
2. No history of non-functional bowel disease(cholangitis, pancreatitis, enteritis, ulcer, bleeding, cancer, etc.)
3. Before participation clinical trial, one who took over-the-count medication affecting GI motility
4. One who takes antibiotics during run-in period (2 wks)
5. One who takes probiotics within 2 wks before experiment
6. Pregnant woman
7. One who disagree on the consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Adequate relief (AR) of IBS pain & discomfort | Weekly (during run-period [2 wks], administarion period [8 wks] and follow-up period [2 wks])
  As the participants answer the question "in the past seven days have you had adequate relief of your irritable bowel syndrome pain and discomfort?" in the form of "Yes" or "No", the effect can be assessed.
Proportion of responders | Once in each period (run-period [2 wks], administarion period [8 wks] and follow-up period [2 wks])
  The proportion of responders who answer "Yes" to more than half of AR questions in each period (>50%)

SECONDARY OUTCOMES:
Daily assessment of bowel function scores | Daily (during run-period [2 wks], administarion period [8 wks] and follow-up period [2 wks])
  1. The patients should write diaries of stool's frequency, consistency and ease of passage
  2. Frequency (number of defecation in a day)
  3. Consistency (judged by Bristol scale)
  4. Ease of passage
Daily assessment of severity of individual symptoms related to defecation | Daily (during run-period [2 wks], administarion period [8 wks] and follow-up period [2 wks])
  Abdominal pain, abdominal discomfort, bloating, flatulence, urgency, mucus in stool and overall symptom would be evaluated through visual analog scale (100mm)
Changes on population of intestinal microbes | Two times in administration period (0 and 8 wks)
  1. To investigate the changes of intestinal microbes before and after experiment, feces should be collected.
  2. The feces will be analyzed by the method of DGGE (denaturing gradient gel electrophoresis - PCR of DNA).
Intestinal permeability test | Two times in administration period (0 and 8 wks)
  In order to evaluate intesinal permeability, the urine should be collected after orally administration of lactulose and mannitol.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Woo Park, KMD, PhD, Principal Investigator — Department of Internal Medicine, College of Oriental Medicine, Kyung Hee University, 1 Hoegi-dong, Dongdaemun-gu, Seoul 130-701, Republic of Korea
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu, South Korea

REFERENCES:
- [Derived] Ko SJ, Ryu B, Kim J, Hong BG, Yeo I, Lee BJ, Lee JM, Park JW. Effect of herbal extract granules combined with probiotic mixture on irritable bowel syndrome with diarrhea: study protocol for a randomized controlled trial. Trials. 2011 Oct 6;12:219. doi: 10.1186/1745-6215-12-219. PMID 21978382
- See also: This is the URL of the site in which the clinical trial will be conducted. — http://www.khnmc.or.kr/